CLINICAL TRIAL: NCT03732586
Title: Effect of Omega-5 Fatty Acid Supplement on Markers of Inflammation and Oxidative Stress in Patients With Severe Alcoholic Hepatitis Treated With Prednisone
Brief Title: Effect of Omega 5 Fatty Acid as an Adyuvant Treatment to Prednisone in Patients With Severe Alcoholic Hepatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Dr. Manuel Gea González (Other Government)
Collaborators: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Jacqueline Cordova-Gallardo, Hepatologist, Hospital General Dr. Manuel Gea González
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hospitalgea
Record Dates: First submitted 2018-10-30; First posted 2018-11-06 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Alcoholic Hepatitis
Keywords: Severe Alcoholic Hepatitis treatment
MeSH Terms: conditions — Hepatitis, Alcoholic

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind clinical trial.
Who Masked: Participant
Masking Description: Subjects will be randomly assigned to one of the two treatments. The randomization is done through a computer generated system. The labelling will be done by a pharmacist or similar. Envelopes with randomization listings will be stored in a secure environment within the Hospital. Blinding should be maintained throughout the study. The randomization code should not be broken during the course of the study unless it is necessary for the safety of the subjects, as judged by the investigator. The date, time and reason for unmasking must be recorded, along with the researcher's signature. The rupture of the study blind will be done once the database has been blocked. The study will be double-blind, which means that neither the patients nor the study site staff will have access to the randomization code until the code is broken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega 5 fatty acid supplement (Experimental): 20 patients will be assigned to traditional treatment with prednisone 40 mg per day plus dietary supplement with omega 5 fatty acid
  Interventions: Dietary Supplement: Omega 5 fatty acid supplement
- PLACEBO (Placebo Comparator): 20 patients will be assigned to traditional treatment (prednisone 40 mg per day) plus placebo
  Interventions: Other: PLACEBO

INTERVENTIONS:
Dietary Supplement: Omega 5 fatty acid supplement — Patients will be randomized to receive traditional treatment (prednisone 40 mg per day) plus omega 5 fatty acid ( 2 capsules of 0.64g per day) for 28 days.
  Arms: Omega 5 fatty acid supplement
Other: PLACEBO — Patients will be randomized to receive the traditional treatment (prednisone 40 mg per day) plus placebo (2 capsules of placebo with identical appereance and size like omega 5 supplement) for 28 days.
  Other Names: placebo capsules
  Arms: PLACEBO

SUMMARY:
In Mexico, alcoholic liver disease is the fourth cause of mortality (INEGI). Patients with severe alcoholic hepatitis have a high mortality at 28 days and 6 months, patients receiving standard therapy with prednisone that are non responders (Lille> 0.45) have a survival of 53.3 ± 5.1 % to 28 days. At present, there is not a completely effective treatment for non responders patients, with a high mortality, so it is necessary to look for other therapeutic strategies.

The omega-5 fatty acid (punicic acid) has been considered a powerful antioxidant, it is an agonist of PPAR gamma, has been shown to reduce lipid peroxidation, and restore levels of antioxidant enzymes such as superoxide dismutase (SOD), catalase and glutathione peroxidase. It has also been shown to inhibit the expression of proinflammatory cytokines (such as IL6, IL8, IL23, IL12 and TNFalpha) through PPAR and modulation delta.

The objective of this study is to evaluate the effect of Omega 5 fatty acid on inflammatory markers and antioxidant-oxidant balance markers in patients with severe alcoholic hepatitis treated with prednisone. HYPOTHESIS. Omega 5 fatty acid being a PPARgamma agonist reduces lipid peroxidation and protein damage, restoring reduced glutathione levels, as well as decreasing proinflammatory cytokines, in patients with Severe Alcoholic Hepatitis treated with prednisone and supplementation with fatty acid Omega 5.

DETAILED DESCRIPTION:
Double-blind clinical trial.

Two groups:

* GROUP A (standard treatment): Prednisone 40 mg a day + Placebo (manufactured by the same laboratory with the same presentation and physical appearance as the nanoemulsifyied pomegranate seed oil rich in Omega 5 fatty acid)
* GROUP B (combined treatment): Prednisone 40 mg per day + nanoemulsifiyied pomegranate seed oil rich in Omega 5 fatty acid (2 capsules of 0.64g each / day).

STUDY UNIVERSE: Patients> 18 years old, indistinct gender, with a diagnosis of severe alcoholic hepatitis.

STUDY POPULATION: Patients with clinical and laboratory diagnosis of alcoholic hepatitis Severe Maddrey score ≥32.

SAMPLE SIZE: Double-blind clinical trial, which will include 20 patients for standard treatment and 20 patients for combined treatment, patients who meet the inclusion criteria will be invited to participate. If they agree to participate (after signing the informed consent), the AUDIT C and CAGE questionnaires will be applied, as well as the measurement of anthropometric values and the taking of 3 blood tubes (2 purple and 1 yellow) for the measurement of cytokines, markers of oxidative stress, lipid peroxidation and protein carbonyls.

The initial evaluation will include liver ultrasound, heart rate, blood pressure, temperature, anthropometric evaluation (weight (kilograms), height (meters), BMI (kg/m2), evaluation of ascites (abdominal circumference), hepatic encephalopathy (West Haven Scale). Alcohol abuse will be assessed using the AUDIT and CAGE score. Start-up laboratories will be carried out: TP, INR, Complete liver function tests (BT, BD, FA, AST, ALT, GGT, Albumin), Seric electrolytes (Na, K, Phosphorus, Magnesium), Creatinine, Blood cytometry (Leukocytes (PMN) ), hemoglobin, VCM, platelets), lipid profile (ColT, HDL, LDL, TGs), ferritin and transferrin saturation, Anti-nuclear antibodies, Anti mithochondrial antibodies, AgHBs, AcHBc, anti HCV, anti HIV. The scrutiny of bacterial infections will be carried out through urine culture, blood cultures and in case of suspicion of SBP (paracenthesis). Child-Pugh score (A5-6, B7-9, C10-12), Maddrey score, MELD, ABIC score, Glasgow score. Chest x-Ray, General Urine Test.

Patients who meet the inclusion criteria, previously described, will be proposed to participate in the study, explaining in detail the procedures as well as the studiesthat will be performed. If they agree to participate, they will proceed to the signature of the informed consent by the patient and their responsible family member. Samples (2 yellow tubes and 2 purple tubes) will be taken for the measurement of cytokines, markers of oxidative stress, lipid peroxidation and protein carbonyls prior to the supply of the supplement vs placebo as well as the start of standard treatment. It will be explained to the patient that these samples will be done in 4 times (at diagnosis, on day 7, 14 and 28), which will be carried out during their hospitalization and follow-up.

Both treatments will be taken for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical and biochemical criteria for severe alcoholic hepatitis (Total bilirubin greater than 5 mg/dl in absence of biliary tract obstruction evidenced by ultrasound)
* history of chronic alcohol intake (greater than 50 g / day for at least 3 months),
* leukocytosis (neutrophilia)
* elevation of transaminases with an aspartate aminotransferase / alanine aminotransferase ratio equal or greater than 2)
* discriminant function greater than 32.

Exclusion Criteria:

* Hepatorenal syndrome (serum creatinine >2.5mg/dl)
* Hepatocellular carcinoma.
* Hepatitis C virus, hepatitis B virus or human immunodeficiency virus infection.
* Cancer, heart disease, neurological or severe neurological.
* Patients taking pentoxifylline, steroids, S-adenosyl L- methionine or N-Acetylcysteine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
30 Day Survival | day 30
  Better survival in patients with omega 5 supplement associated to prednisone

SECONDARY OUTCOMES:
Rate of reponse to steroids at day 7 | day 7
  To describe the response to steroids (Lille score) at 7 days of treatment in patients with severe alcoholic hepatitis with combined treatment (Omega 5 and steroids) compared to standard treatment. (Lille response describe a below of 0.45)
Malondialdehyde serum levels | basal, day 7, day 14 and day 28
  To determine the serum concentrations of lipid peroxidation molecules (malondialdehyde (MDA expressed in mM) in patients with severe alcoholic hepatitis treated with prednisone compare to those treated with prednisona and omega5.
Oxidative Stress molecules serum levels | basal, day 7, day 14 and day 28
  To assess changes in oxidative stress markers (Oxidative glutation and reduced glutation expressed in mM) in patients with severe alcoholic hepatitis treated with prednisone compared to those treated with prednisone and omega 5.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Cordova-Gallardo, MD, Principal Investigator — Hospital General Dr. Manuel Gea Gonzalez; Gabriela Gutierrez-Reyes, DSc, Principal Investigator — Universidad Autonoma de México
Locations (2):
- Mexico (2):
  - Laboratorio de Higado, Pancreas y Motilidad Intestinal. UNIVERSIDAD AUTONOMA DE MEXICO, Mexico City, Cuauhtemoc
  - Hospital General Dr. Manuel Gea Gonzalez, Mexico City, Tlalpan

IPD SHARING:
Plan to Share IPD: No
The results will be shared in international medical meetings

REFERENCES:
- [Background] European Association for the Study of Liver. EASL clinical practical guidelines: management of alcoholic liver disease. J Hepatol. 2012 Aug;57(2):399-420. doi: 10.1016/j.jhep.2012.04.004. Epub 2012 May 26. No abstract available. PMID 22633836
- [Background] Mendez-Sanchez N, Villa AR, Chavez-Tapia NC, Ponciano-Rodriguez G, Almeda-Valdes P, Gonzalez D, Uribe M. Trends in liver disease prevalence in Mexico from 2005 to 2050 through mortality data. Ann Hepatol. 2005 Jan-Mar;4(1):52-5. PMID 15798662
- [Background] Amini M, Runyon BA. Alcoholic hepatitis 2010: a clinician's guide to diagnosis and therapy. World J Gastroenterol. 2010 Oct 21;16(39):4905-12. doi: 10.3748/wjg.v16.i39.4905. PMID 20954276
- [Background] Lucey MR, Mathurin P, Morgan TR. Alcoholic hepatitis. N Engl J Med. 2009 Jun 25;360(26):2758-69. doi: 10.1056/NEJMra0805786. No abstract available. PMID 19553649
- [Background] Nguyen-Khac E, Thevenot T, Piquet MA, Benferhat S, Goria O, Chatelain D, Tramier B, Dewaele F, Ghrib S, Rudler M, Carbonell N, Tossou H, Bental A, Bernard-Chabert B, Dupas JL; AAH-NAC Study Group. Glucocorticoids plus N-acetylcysteine in severe alcoholic hepatitis. N Engl J Med. 2011 Nov 10;365(19):1781-9. doi: 10.1056/NEJMoa1101214. PMID 22070475
- [Background] Thursz MR, Richardson P, Allison M, Austin A, Bowers M, Day CP, Downs N, Gleeson D, MacGilchrist A, Grant A, Hood S, Masson S, McCune A, Mellor J, O'Grady J, Patch D, Ratcliffe I, Roderick P, Stanton L, Vergis N, Wright M, Ryder S, Forrest EH; STOPAH Trial. Prednisolone or pentoxifylline for alcoholic hepatitis. N Engl J Med. 2015 Apr 23;372(17):1619-28. doi: 10.1056/NEJMoa1412278. PMID 25901427
- [Background] Basra G, Basra S, Parupudi S. Symptoms and signs of acute alcoholic hepatitis. World J Hepatol. 2011 May 27;3(5):118-20. doi: 10.4254/wjh.v3.i5.118. PMID 21731904
- [Background] Sass DA, Shaikh OS. Alcoholic hepatitis. Clin Liver Dis. 2006 May;10(2):219-37, vii. doi: 10.1016/j.cld.2006.05.011. PMID 16971259
- [Background] Ambade A, Mandrekar P. Oxidative stress and inflammation: essential partners in alcoholic liver disease. Int J Hepatol. 2012;2012:853175. doi: 10.1155/2012/853175. Epub 2012 Mar 1. PMID 22500241
- [Background] Lefkowitch JH. Morphology of alcoholic liver disease. Clin Liver Dis. 2005 Feb;9(1):37-53. doi: 10.1016/j.cld.2004.11.001. PMID 15763228
- [Background] Dugum MF, McCullough AJ. Acute Alcoholic Hepatitis, the Clinical Aspects. Clin Liver Dis. 2016 Aug;20(3):499-508. doi: 10.1016/j.cld.2016.02.008. Epub 2016 May 14. PMID 27373612
- [Background] Cohen SM, Ahn J. Review article: the diagnosis and management of alcoholic hepatitis. Aliment Pharmacol Ther. 2009 Jul;30(1):3-13. doi: 10.1111/j.1365-2036.2009.04002.x. Epub 2009 Mar 26. PMID 19416132
- [Background] Gholam PM. Prognosis and Prognostic Scoring Models for Alcoholic Liver Disease and Acute Alcoholic Hepatitis. Clin Liver Dis. 2016 Aug;20(3):491-7. doi: 10.1016/j.cld.2016.02.007. Epub 2016 May 14. PMID 27373611
- [Background] Sheth M, Riggs M, Patel T. Utility of the Mayo End-Stage Liver Disease (MELD) score in assessing prognosis of patients with alcoholic hepatitis. BMC Gastroenterol. 2002;2:2. doi: 10.1186/1471-230x-2-2. Epub 2002 Jan 22. PMID 11835693
- [Background] Dominguez M, Rincon D, Abraldes JG, Miquel R, Colmenero J, Bellot P, Garcia-Pagan JC, Fernandez R, Moreno M, Banares R, Arroyo V, Caballeria J, Gines P, Bataller R. A new scoring system for prognostic stratification of patients with alcoholic hepatitis. Am J Gastroenterol. 2008 Nov;103(11):2747-56. doi: 10.1111/j.1572-0241.2008.02104.x. Epub 2008 Aug 21. PMID 18721242
- [Background] Higuera-de la Tijera MF, Perez-Hernandez JL, Serralde-Zuniga AE, Servin-Caamano AI, Cruz-Palacios A, Bernal-Sahagun F, Salas-Gordillo F. [Three prognostic utility scales to determine early mortality in patients with alcoholic hepatitis in the General Hospital of Mexico]. Rev Gastroenterol Mex. 2010;75(3):281-6. Spanish. PMID 20959177
- [Background] Altamirano J, Higuera-de laTijera F, Duarte-Rojo A, Martinez-Vazquez MA, Abraldes JG, Herrera-Jimenez LE, Michelena J, Zapata L, Perez-Hernandez J, Torre A, Gonzales-Gonzalez JA, Cardenas A, Dominguez M, Arroyo V, Gines P, Caballeria J, Bataller R. The amount of alcohol consumption negatively impacts short-term mortality in Mexican patients with alcoholic hepatitis. Am J Gastroenterol. 2011 Aug;106(8):1472-80. doi: 10.1038/ajg.2011.141. Epub 2011 May 10. PMID 21556041
- [Background] Higuera-de la Tijera MF, Perez-Hernandez JL, Servin-Caamano AL, Serralde-Zuniga AE, Cruz-Palacios A. [The amount of alcohol intake, upper gastrointestinal bleeding, acute renal failure and hepatic encephalopathy as the risk factors implied in the increase of patients with alcoholic hepatitis]. Rev Gastroenterol Mex. 2009 Oct-Dec;74(4):306-13. Spanish. PMID 20423759
- [Background] Louvet A, Wartel F, Castel H, Dharancy S, Hollebecque A, Canva-Delcambre V, Deltenre P, Mathurin P. Infection in patients with severe alcoholic hepatitis treated with steroids: early response to therapy is the key factor. Gastroenterology. 2009 Aug;137(2):541-8. doi: 10.1053/j.gastro.2009.04.062. Epub 2009 May 13. PMID 19445945
- [Background] Louvet A, Naveau S, Abdelnour M, Ramond MJ, Diaz E, Fartoux L, Dharancy S, Texier F, Hollebecque A, Serfaty L, Boleslawski E, Deltenre P, Canva V, Pruvot FR, Mathurin P. The Lille model: a new tool for therapeutic strategy in patients with severe alcoholic hepatitis treated with steroids. Hepatology. 2007 Jun;45(6):1348-54. doi: 10.1002/hep.21607. PMID 17518367
- [Background] Phillips PK, Lucey MR. Acute Alcoholic Hepatitis: Therapy. Clin Liver Dis. 2016 Aug;20(3):509-19. doi: 10.1016/j.cld.2016.02.015. Epub 2016 May 31. PMID 27373613
- [Background] Higuera-de la Tijera F, Servin-Caamano AI, Serralde-Zuniga AE, Cruz-Herrera J, Perez-Torres E, Abdo-Francis JM, Salas-Gordillo F, Perez-Hernandez JL. Metadoxine improves the three- and six-month survival rates in patients with severe alcoholic hepatitis. World J Gastroenterol. 2015 Apr 28;21(16):4975-85. doi: 10.3748/wjg.v21.i16.4975. PMID 25945012
- [Background] Mathurin P, O'Grady J, Carithers RL, Phillips M, Louvet A, Mendenhall CL, Ramond MJ, Naveau S, Maddrey WC, Morgan TR. Corticosteroids improve short-term survival in patients with severe alcoholic hepatitis: meta-analysis of individual patient data. Gut. 2011 Feb;60(2):255-60. doi: 10.1136/gut.2010.224097. Epub 2010 Oct 12. PMID 20940288
- [Result] Bihamta M, Hosseini A, Ghorbani A, Boroushaki MT. Protective effect of pomegranate seed oil against H2O2 -induced oxidative stress in cardiomyocytes. Avicenna J Phytomed. 2017 Jan-Feb;7(1):46-53. PMID 28265546
- [Result] Boroushaki MT, Hosseini A, Dolati K, Mollazadeh H, Rajabian A. PROTECTIVE EFFECT OF POMEGRANATE SEED OIL AGAINST MERCURIC CHLORIDE-INDUCED HEPATOTOXICITY IN RAT. Acta Pol Pharm. 2016 Jul;73(4):991-997. PMID 29648725
- [Result] Boroushaki MT, Rajabian A, Farzadnia M, Hoseini A, Poorlashkari M, Taghavi A, Dolati K, Bazmandegan G. Protective effect of pomegranate seed oil against cisplatin-induced nephrotoxicity in rat. Ren Fail. 2015;37(8):1338-43. doi: 10.3109/0886022X.2015.1073496. Epub 2015 Aug 14. PMID 26288026
- [Result] Nematbakhsh M. Cisplatin and herbal antioxidants: protective effect of pomegranate seed oil against cisplatin-induced nephrotoxicity in rat. Ren Fail. 2016;38(2):344-5. doi: 10.3109/0886022X.2015.1127740. Epub 2015 Dec 27. No abstract available. PMID 26707061
- [Result] Boroushaki MT, Mollazadeh H, Rajabian A, Dolati K, Hoseini A, Paseban M, Farzadnia M. Protective effect of pomegranate seed oil against mercuric chloride-induced nephrotoxicity in rat. Ren Fail. 2014 Nov;36(10):1581-6. doi: 10.3109/0886022X.2014.949770. Epub 2014 Aug 26. PMID 25154291
- [Result] Boroushaki MT, Rajabian A, Farzadnia M, Hoseini A, Poorlashkari M, Taghavi A, Dolati K, Bazmandegan G. Protective effect of pomegranate seed oil against cisplatin-induced nephrotoxicity in rat. Ren Fail. 2015 Aug 14:1-6. Online ahead of print. PMID 26275112
- [Result] Mollazadeh H, Sadeghnia HR, Hoseini A, Farzadnia M, Boroushaki MT. Effects of pomegranate seed oil on oxidative stress markers, serum biochemical parameters and pathological findings in kidney and heart of streptozotocin-induced diabetic rats. Ren Fail. 2016 Sep;38(8):1256-66. doi: 10.1080/0886022X.2016.1207053. Epub 2016 Jul 25. PMID 27453190
- [Result] Boroushaki MT, Arshadi D, Jalili-Rasti H, Asadpour E, Hosseini A. Protective effect of pomegranate seed oil against acute toxicity of diazinon in rat kidney. Iran J Pharm Res. 2013 Fall;12(4):821-7. PMID 24523762
- [Result] Shaban NZ, El-Kersh MA, El-Rashidy FH, Habashy NH. Protective role of Punica granatum (pomegranate) peel and seed oil extracts on diethylnitrosamine and phenobarbital-induced hepatic injury in male rats. Food Chem. 2013 Dec 1;141(3):1587-96. doi: 10.1016/j.foodchem.2013.04.134. Epub 2013 May 23. PMID 23870864
- [Result] Coursodon-Boyiddle CF, Snarrenberg CL, Adkins-Rieck CK, Bassaganya-Riera J, Hontecillas R, Lawrence P, Brenna JT, Jouni ZE, Dvorak B. Pomegranate seed oil reduces intestinal damage in a rat model of necrotizing enterocolitis. Am J Physiol Gastrointest Liver Physiol. 2012 Sep 15;303(6):G744-51. doi: 10.1152/ajpgi.00248.2012. Epub 2012 Jul 19. PMID 22821948
- [Result] Mollazadeh H, Boroushaki MT, Soukhtanloo M, Afshari AR, Vahedi MM. Effects of pomegranate seed oil on oxidant/antioxidant balance in heart and kidney homogenates and mitochondria of diabetic rats and high glucose-treated H9c2 cell line. Avicenna J Phytomed. 2017 Jul-Aug;7(4):317-333. PMID 28884082
- [Result] Cao Y, Yang L, Gao HL, Chen JN, Chen ZY, Ren QS. Re-characterization of three conjugated linolenic acid isomers by GC-MS and NMR. Chem Phys Lipids. 2007 Feb;145(2):128-33. doi: 10.1016/j.chemphyslip.2006.11.005. Epub 2006 Dec 1. PMID 17204261
- [Result] Baccarin T, Mitjans M, Ramos D, Lemos-Senna E, Vinardell MP. Photoprotection by Punica granatum seed oil nanoemulsion entrapping polyphenol-rich ethyl acetate fraction against UVB-induced DNA damage in human keratinocyte (HaCaT) cell line. J Photochem Photobiol B. 2015 Dec;153:127-36. doi: 10.1016/j.jphotobiol.2015.09.005. Epub 2015 Sep 4. PMID 26406978
- [Result] Mirmiran P, Fazeli MR, Asghari G, Shafiee A, Azizi F. Effect of pomegranate seed oil on hyperlipidaemic subjects: a double-blind placebo-controlled clinical trial. Br J Nutr. 2010 Aug;104(3):402-6. doi: 10.1017/S0007114510000504. Epub 2010 Mar 25. PMID 20334708
- [Result] Viladomiu M, Hontecillas R, Lu P, Bassaganya-Riera J. Preventive and prophylactic mechanisms of action of pomegranate bioactive constituents. Evid Based Complement Alternat Med. 2013;2013:789764. doi: 10.1155/2013/789764. Epub 2013 Apr 30. PMID 23737845
- [Result] Arao K, Yotsumoto H, Han SY, Nagao K, Yanagita T. The 9cis,11trans,13cis isomer of conjugated linolenic acid reduces apolipoprotein B100 secretion and triacylglycerol synthesis in HepG2 cells. Biosci Biotechnol Biochem. 2004 Dec;68(12):2643-5. doi: 10.1271/bbb.68.2643. PMID 15618643
- [Result] Baccarin T, Mitjans M, Lemos-Senna E, Vinardell MP. Protection against oxidative damage in human erythrocytes and preliminary photosafety assessment of Punica granatum seed oil nanoemulsions entrapping polyphenol-rich ethyl acetate fraction. Toxicol In Vitro. 2015 Dec 25;30(1 Pt B):421-8. doi: 10.1016/j.tiv.2015.09.020. Epub 2015 Sep 25. PMID 26407526
- [Result] Mizrahi M, Friedman-Levi Y, Larush L, Frid K, Binyamin O, Dori D, Fainstein N, Ovadia H, Ben-Hur T, Magdassi S, Gabizon R. Pomegranate seed oil nanoemulsions for the prevention and treatment of neurodegenerative diseases: the case of genetic CJD. Nanomedicine. 2014 Aug;10(6):1353-63. doi: 10.1016/j.nano.2014.03.015. Epub 2014 Apr 2. PMID 24704590
- [Result] Harzallah A, Hammami M, Kepczynska MA, Hislop DC, Arch JR, Cawthorne MA, Zaibi MS. Comparison of potential preventive effects of pomegranate flower, peel and seed oil on insulin resistance and inflammation in high-fat and high-sucrose diet-induced obesity mice model. Arch Physiol Biochem. 2016;122(2):75-87. doi: 10.3109/13813455.2016.1148053. Epub 2016 Feb 26. PMID 26822470
- [Result] Miranda J, Arias N, Fernandez-Quintela A, del Puy Portillo M. Are conjugated linolenic acid isomers an alternative to conjugated linoleic acid isomers in obesity prevention? Endocrinol Nutr. 2014 Apr;61(4):209-19. doi: 10.1016/j.endonu.2013.04.016. Epub 2013 Sep 10. English, Spanish. PMID 24029409
- [Result] Holic R, Xu Y, Caldo KMP, Singer SD, Field CJ, Weselake RJ, Chen G. Bioactivity and biotechnological production of punicic acid. Appl Microbiol Biotechnol. 2018 Apr;102(8):3537-3549. doi: 10.1007/s00253-018-8883-y. Epub 2018 Mar 3. PMID 29502183